CLINICAL TRIAL: NCT01438242
Title: An Open Label Study of the Genecept™ Assay to Evaluate Efficacy of Using Assay Guided Treatment in Outpatient Adults With Treatment Resistant Depression
Brief Title: An Open Label Study of the Genecept™ Assay in Treatment Resistant Depression
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Genomind, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AT1
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Major Depressive Disorder
Keywords: Major; Depressive; Disorder; Depression; Treatment Resistant
MeSH Terms: conditions — Depressive Disorder, Major; Disease; Depression | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assay Guided Treatment - Genecept Asay (Experimental): Subjects donate DNA sample for genetic testing and treatment decisions take genetic results into account. Genetic analysis is performed using the Genecept Assay, a genetic test which analyzes seven pharmacodynamic and three pharmacokinetic genes important in psychiatric disorders
  Interventions: Device: Genecept Assay
- Clinician's utilizing Assay Guided Treatment in Psychiatry (Experimental): Prescribing clinicians responsible for the treatment of patients age 18 and older with a primary diagnosis of Major Depressive Disorder or Generalized Anxiety disorder, and for whom the Genecept Assay has been utilized to perform genetic testing.
  Interventions: Device: Genecept Assay

INTERVENTIONS:
Device: Genecept Assay — Genetic test which analyzes seven pharmacodynamic and three pharmacokinetic genes important in psychiatric disorders
  Other Names: Genetic Test

SUMMARY:
The purpose of this study is to examine the potential impact of the assay in terms of depression severity as measured by change in Clinical Global Impressions (CGI) scale at 3 months.

DETAILED DESCRIPTION:
Genomind is sponsoring an open label study of Assay Guided Treatment (AGT) using the Genecept Assay in adult outpatients with Treatment Resistant Major Depressive Disorder. The Genecept Assay is a Clinical Laboratory Improvement Amendments (CLIA) laboratory validated test being researched to determine if having information about genetic variations impacts patient outcomes.

The proposed investigation will examine the potential impact of the Assay in terms of depression severity as measured by change in CGI scale at 3 months. Secondary measures will assess change in Quick Inventory of Depressive Symptoms (QIDS-SR), Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) and Zung self-rated anxiety scales at 3 months. Additional measures include change in clinician treatment and diagnosis decisions and impact on mediation side effects using the Udvalg for Kliniske Undersøgelser Side Effect Rating Scale (UKU). Participant data will be compared to a matched control cohort to assess the impact of the use of the Genecept Assay on medication adherence and total claims.

Patients with a diagnosis of non-psychotic Major Depressive Disorder will be identified. These patients and their treating clinicians will be recruited. The present study proposes to enroll 1. Subjects (patients who are identified as eligible) and 2. Clinician study participants (clinicians who are identified as responsible for the care of eligible patients). This study will involve the collection of responses from both Subjects and clinician study participants with the intention of correlating this information to Subject genetic data.

Potential subjects and study participants will consent electronically on a secure study portal. Patients and Clinicians must both consent to participate in order to proceed in the study. After both subjects and clinician study participants have consent to participate, they will each be asked to complete an electronic baseline survey. Once the baseline survey is completed, the clinician will receive the Genecept Assay by mail and will then supervise collection of a saliva DNA sample during a routine office visit.

At baseline, month 1 and month 3, patient Subjects will be prompted to complete surveys which include questions about their psychiatric symptoms, quality of life and medication side effects. The 3 month patient assessment will also include a satisfaction questionnaire.

At baseline, clinician study participants will be prompted to complete a brief survey containing questions about the patient's psychiatric history and severity of illness, current treatment regimen and the treatment intentions of the clinician prior to receiving genetic results. After receiving the results of the Assay, clinician study participants will again be prompted to complete an online study survey containing questions related to the impact of the Genecept Assay on treatment and diagnosis decisions. The subject will continue with treatment as determined by the clinician study participant. At 3 months from baseline, clinician study participants will again be asked to complete an online survey with additional questions related to subsequent changes to the patient's treatment regimen and illness severity since receiving/implementing the results of the Assay.

ELIGIBILITY:
Subjects:

Inclusion Criteria:

* Age 18-65 years
* Ability to complete electronic informed consent

Includes:

* access to appropriate technology (i.e. internet-connected device, internet connection),
* cognitively competent

  * Eligible participants will have one or more of the following diagnoses for 12 months or longer: 296.2x, 296.3x
  * Must have had self-insured Aetna Behavioral Health, Medical, and Pharmacy benefits for that 12-month period.
  * QIDS-SR score of at least 10 (i.e., moderate depression) at initial visit
  * Must have had an initial prescription plus two refills of two antidepressants from different GPI4 levels.
  * Must have access to the secure web-portal to complete self-assessments

Exclusion Criteria:

* Clinician selected in conjunction with the patient chooses not to participate
* Psychotic features in the current episode, based upon clinical assessment
* Inpatient behavioral health hospitalization within six months prior to the study
* Four or more failed pharmacologic interventions in the current major depressive episode [response rates for these Subjects is likely to be extremely low and would require a substantially larger-scale study to identify treatment effects]
* Current substance use disorder assessed as being of a severity that requires inpatient or outpatient detoxification
* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception
* Women who are breastfeeding
* Serious suicide or homicide risk, as assessed by evaluating clinician
* Unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease, based on review of medical history, physical examination, and screening laboratory tests
* Patients who have taken an investigational psychotropic drug within the last three months

Clinician Study Participants:

Inclusion Criteria :

* Treating clinician for potential Patient subjects identified for the study
* Valid NPI number
* Signed electronic informed consent

Exclusion Criteria:

* Inability to complete online surveys
* Patient selected in conjunction with the clinician chooses not to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 3 Months
  To determine the efficacy of assay-guided treatment (AGT) in terms of illness severity as measured by change from baseline in Clinical Global Impressions (CGI) scale at 3 months.

SECONDARY OUTCOMES:
Efficacy | 3 months
  To determine the efficacy of assay-guided treatment (AGT) in terms of illness severity as measured by change from baseline in Quick Inventory of Depressive Symptoms (QIDS-SR1), Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) and Zung self-rated anxiety scales at 3 months.
Medication Adherence | 3 months
  To compare medication adherence between Patient subjects and matched control cohort
Resource Utilization | 3 months
  To determine the comparative effectiveness of AGT versus Treatment as Usual (TAU) in a matched control cohort in outpatient management of nonpsychotic Major Depressive Disorder patients with treatment resistant depression, as measured by total claims.
Impact of Specific Genetic Variants | 3 months
  1. To explore genetic variants within the patient population and identify subgroups for whom pharmacogenetic testing is particularly informative
  2. To determine which specific results of pharmacogenetic testing have the most impact on clinician behavior
Side Effects | 3 months
  To explore genetic variants in relationship to classes of medications and treatment response as measured by CGI and QIDs, and change in reported adverse events using the UKU (The Udvalg for Kliniske Undersøgelser Side Effect Rating Scale.)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Harris, MD, PhD, Principal Investigator — Rho, Inc.
Locations (1):
- Genomind, LLC, Chalfont, Pennsylvania, United States